CLINICAL TRIAL: NCT01674829
Title: A Phase I/IIa, Open-Label, Single-Center, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (MA09-hRPE) Cells in Patients With Advanced Dry Age-related Macular Degeneration(AMD)
Brief Title: A PhaseI/IIa Study to Determine the Safety and Tolerability of MA09-hRPE Cells in Patients With Advanced Dry AMD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: CHABiotech CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHA CTP 1101
Record Dates: First submitted 2012-08-22; First posted 2012-08-29 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Dry Age Related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Biological: MA09-hRPE Cellular therapy Cohort 1 Dose 1
  Interventions: Biological: MA09-hRPE
- Cohort 2 (Experimental): Biological: MA09-hRPE Cellular therapy Cohort 2 Dose 2
  Interventions: Biological: MA09-hRPE
- Cohort 3 (Experimental): Biological: MA09-hRPE Cellular therapy Cohort 3 Dose 3
  Interventions: Biological: MA09-hRPE
- Cohort 4 (Experimental): Biological: MA09-hRPE Cellular therapy Cohort 4 Dose 4
  Interventions: Biological: MA09-hRPE

INTERVENTIONS:
Biological: MA09-hRPE — Transplantation of MA09-hRPE cells accoding to the assigned dose group

SUMMARY:
To evaluate the safety and tolerability of MA09-hRPE cellular therapy in patients with advanced dry AMD To evaluate the safety of the surgical procedures when used to implant MA09-hRPE cells To assess the number of hRPE cells to be transplanted in future studies To evaluate on an exploratory basis potential efficacy endpoints to be used in future studies of MA09-hRPE cellular therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over 55 years of age. Patient should be in sufficiently good health to reasonably expect survival for at least four years after treatment
* Clinical findings consistent with advanced dry AMD
* GA defined as attenuation or loss of RPE as observed by biomicroscopy, OCT, and FA.
* No evidence of current or prior choroidal neovascularization in the treated eye
* The visual acuity (BCVA) of the eye to receive the transplant found to be eligible for trial based on study protocol
* Electrophysiological findings consistent with advanced dry AMD.
* Medically suitable to undergo vitrectomy and subretinal injection.
* Medically suitable for general anesthesia or waking sedation, if needed.
* Medically suitable for transplantation of an embryonic stem cell line

Exclusion Criteria:

* Presence of active or inactive CNV in the eye to be treated.
* Presence or history of retinal dystrophy, retinitis pigmentosa, chorioretinitis, central serious choroidopathy, diabetic retinopathy or other retinal vascular or degenerative disease other than ARMD.
* History of optic neuropathy.
* Macular atrophy due to causes other than AMD.
* Presence of glaucomatous optic neuropathy in the study eye, uncontrolled IOP, or use of two or more agents to control IOP (acetazolamide, beta blocker, alpha-1-agonist, prostaglandins, anhydrous carbonic inhibitors)
* Cataract of sufficient severity likely to necessitate surgical extraction within 1 year.
* History of retinal detachment repair in the study eye.
* History of myocardial infarction in previous 12 months.
* History of diabetes mellitus.
* History of cognitive impairments or dementia which may impact the patients ability participate in the informed consent process and to appropriately complete evaluations.
* Any immunodeficiency.
* Any abnormalities in laboratory test result.
* Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV.
* Current participation in any other clinical trial.
* Participation within previous 6 months in any clinical trial of a drug by ocular or systemic administration.
* Any other sight-threatening ocular disease.
* Ocular lens removal within previous 3 months.
* Ocular surgery in the study eye in the previous 3 months
* If female, pregnancy or lactation.
* Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Safety of hESC derived RPE cells | 12 months
  The transplantation of hESC-derived RPE cells MA09-hRPE will be considered safe in the absence of:
  1. Any grade 2 (NCI grading system) or greater adverse event related to the cell product
  2. Any evidence that the cells are contaminated with an infectious agent
  3. Any evidence that the cells show tumorigenic potential

SECONDARY OUTCOMES:
exploratory evaluations for potential efficacy endpoints | 12months
  Secondary endpoints will be evaluated as exploratory evaluations for potential efficacy endpoints.
  * Change in the mean of BCVA
  * Autofluorescense photography
  * Reading speed
  Evidence of successful engraftment will consist of:
  * Structural evidence (OCT imaging, fluorescein angiography, slitlamp examination with fundus photography) that cells have been implanted in the correct location
  * Electroretinographic evidence (mfERG) showing enhanced activity in the implant location

CONTACTS AND LOCATIONS:
Overall Officials: Yeong je Seong, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea